CLINICAL TRIAL: NCT02206776
Title: Randomized Controlled Trial of Intranasal Ketamine vs. Intranasal Midazolam in Individuals With Obsessive Compulsive Disorder (OCD)
Brief Title: Randomized Controlled Trial of Intranasal Ketamine vs. Intranasal Midazolam in Individuals With OCD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: poor tolerability and low enrollment rate
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: #6952
Record Dates: First submitted 2014-07-31; First posted 2014-08-01 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2017-05-03 (Actual); Status verified 2017-03

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: OCD
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Midazolam (Placebo Comparator): A single dose of intranasal midazolam up to 4 mg
  Interventions: Drug: Intranasal Midazolam
- Ketamine (Experimental): A single dose of intranasal ketamine up to 50 mg
  Interventions: Drug: Intranasal Ketamine

INTERVENTIONS:
Drug: Intranasal Ketamine — A single dose of intranasal ketamine up to 50 mg
  Other Names: Ketamine Hydrochloride
  Arms: Ketamine
Drug: Intranasal Midazolam — A single dose of intranasal Midazolam up to 4 mg
  Arms: Midazolam

SUMMARY:
Obsessive-compulsive disorder (OCD) is a common illness that causes significant distress and impairment. Currently, serotonin reuptake inhibitors (SRIs) are the only medications that are FDA-approved to treat OCD. Unfortunately, SRIs can take a long time to work (2-3 months), and even then they usually only partially reduce OCD symptoms. The present study, will test if intranasal ketamine is feasible to use and can reduce OCD symptoms significantly more than a comparison medication called midazolam. Therefore, you may or may not receive ketamine as part of this study. Results from this study will allow doctors and researchers to better understand if you and others with OCD may respond to this class of medications.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55
* Physically healthy and not currently pregnant
* Primary diagnosis of OCD
* Sufficient severity of symptoms
* For all patients on medications, medications dose must be stable for at least 6 weeks prior to enrollment. Must discuss with Dr. current medications and doses.
* Able to provide consent

Exclusion Criteria:

* First degree relative with schizophrenia
* Psychiatric conditions that would make participation unsafe determined by study doctor
* Female patients who are either pregnant or nursing
* Planning to start EX/RP during the period of the study or those who have completed an adequate dose of EX/RP (defined as 8 or more sessions within 2 months) within 8 weeks prior to enrollment.
* Nasal obstruction or history of nasal surgery
* Currently on psychotropic medication or other medication likely to interact with the glutamate system
* Medical conditions that make participation unsafe
* Allergy or intolerance to ketamine or midazolam

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2014-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn I Rodriguez, M.D., Ph.D., Principal Investigator — Stanford University
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://columbia-ocd.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Midazolam | Ketamine
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Midazolam | Ketamine | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 20 (0) | 36 (0) | 28 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Met and Exceeded Response Criteria of Yale-Brown Obsessive-Compulsive Scale.
Description: Patients given YBOCS (Yale Brown Obsessive-Compulsive Scale), a gold standard measure of obsessions and compulsions. For the YBOCS the minimum units are 0 and Maximum units on the total scale are 40. The higher the number on the YBOCS, the more severe the symptoms. Response was defined as at least a 35% reduction on the YBOCS.
Time Frame: Baseline and 1 Week
Measure: Count of Participants; unit: Participants
Arm/Group | Midazolam | Ketamine
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Midazolam | Ketamine
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Midazolam (N=1) | Ketamine (N=1)
perceptual changes (e.g. feeling as if body changed in size) (Psychiatric disorders) | 1 (1) | 1 (1)
headache (Nervous system disorders) | 1 (1) | 0 (0)
lighheadedness (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No